CLINICAL TRIAL: NCT00578864
Title: PEPI: Protracted Etoposide in a Phase II Upfront Window for Induction Therapy for High Risk Neuroblastoma
Brief Title: Protracted Etoposide During Induction Therapy for High Risk Neuroblastoma
Acronym: PEPI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Heidi Russell, Principal investigator, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H20255; PEPI (Other: BCM); NCT00600132 (obsolete NCT alias)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2012-11-06 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Etoposide; Cisplatin; Adriamycin; Cyclophosphamide; Cytoxan
MeSH Terms: conditions — Neuroblastoma | interventions — Doxorubicin; Cisplatin; Cyclophosphamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Protracted Oral Etoposide (Experimental): Protracted oral etoposide for cycles 1, 2 and 4 of induction. Etoposide will be given in combination with IV cisplatin (a standard of care agent). If a subject does not respond after cycle 2, cycle 4 will be bolus etoposide in combination with IV cisplatin.
  All patients will receive Adriamycin and cyclophosphamide for cycle 3 and 5 as a standard of care.
  Interventions: Drug: Protracted Oral Etoposide; Drug: Doxorubicin; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Mesna; Drug: Hematopoietic Factor; Procedure: Primary tumor resection
- IV Bolus Etoposide (Active Comparator): IV bolus etoposide in combination with IV cisplatin will be given for cycles 1,2, and 4 of induction chemotherapy for patients who are not eligible for the experimental arm (e.g.require emergent treatment)
  All patients will receive Adriamycin and cyclophosphamide for cycle 3 and 5 as a standard of care.
  Interventions: Drug: Doxorubicin; Drug: IV Bolus Etoposide; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Mesna; Drug: Hematopoietic Factor; Procedure: Primary tumor resection

INTERVENTIONS:
Drug: Protracted Oral Etoposide — Cisplatin with Oral Protracted Etoposide for cycles 1, 2 and 4
  Day 1 - 5
  * Hour 0: Etoposide 50 mg/m2 po daily
  * Hours 1 to 7: Cisplatin 40 mg/m2
  Day 6 - 14
  * Etoposide 50 mg/m2 po once daily
  Arms: Protracted Oral Etoposide
Drug: Doxorubicin — Given together with cyclophosphamide for cycle 3 and 5 of induction chemotherapy Day 1 and 2
  * Hours 0 to 6: Cyclophosphamide 2000 mg/m2 (67 mg/kg if < 12 kg) with Mesna 400 mg/m2 (13 mg/kg if < 12 kg) in D5½NS 600 mL/m2 IV over 6 hours to run at 100 mL/m2/hr
  * Hours 6 to 6.25: Doxorubicin 37.5 mg/m2 (1.25 mg/kg if < 12 kg) IV over 15 minutes
Drug: IV Bolus Etoposide — Cisplatin with Bolus IV Etoposide
  Day 1
  Hours 0 to 6: Cisplatin 40 mg/m2
  Days 2, 3, 4:
  Hours 0 to 1: Etoposide 200 mg/m2 Hours 1 to 7: Cisplatin 40 mg/m2
  Day 5:
  Hours 0 to 6: Cisplatin 40 mg/m2
  Arms: IV Bolus Etoposide
Drug: Cisplatin — Cycle 1, 2, and 4
Drug: Cyclophosphamide — Cycle 3 and 5 with doxorubicin
Drug: Mesna — Standard weight-based dosing with cyclophosphamide
Drug: Hematopoietic Factor — Standard weight-based dosing after cycle 3 and 5 and if needed for neutropenic recovery after cycles 1,2 and 4
Procedure: Primary tumor resection — Resection of primary tumor after cycle 3, 4, or 5 as clinically appropriate

SUMMARY:
High-risk neuroblastoma is an aggressive childhood cancer that shows up as a lump or mass in the belly or around the spinal cord in the chest, neck, or pelvis. Often the tumor has spread around the body to the bones or to the soft center of the bone, called the bone marrow. High-risk neuroblastoma often responds to treatment at first, but it frequently comes back and may be even more difficult to treat.

Chemotherapy (drug treatments for cancer) is usually given at high doses in short bursts (3 to 5 days) followed by a few weeks of rest and recovery. This burst and recovery is called a "cycle" and usually takes about 21 days. Some scientists and physicians have tried to give chemotherapy at lower doses for more days, called "metronomic" chemotherapy. This method of giving chemotherapy has been used to treat neuroblastoma that has failed more standard types of treatment (relapsed neuroblastoma) and has shown some promise for those patients. One of the reasons it may work is by killing the blood vessels that feed the tumor as well as killing tumor cells themselves (the way that burst chemotherapy works). We think that giving a burst of chemotherapy together with metronomic therapy may kill the tumor while decreasing the side effects that we have seen in the past.

Treatment for high risk neuroblastoma usually occurs in 3 stages: induction, consolidation, and maintenance. During the induction phase, patients will receive chemotherapy and possibly more surgery to get rid of most of the tumor cells. Most of the chemotherapy drugs during induction will be given in the standard burst method. One of the chemotherapy drugs, etoposide, will be given in lower, metronomic doses. The doctors will study how the tumors respond and the side effects patients have. After induction most childrens' tumors will have disappeared, also called remission. These children will receive the second stage of treatment called consolidation. During this stage, subjects will receive radiation treatments to the tumor and then higher doses of chemotherapy. Because of the side effects of the high doses of chemotherapy, we will collect and store some special blood cells (called hematopoietic stem cells) early in treatment and keep them frozen. After the high doses of chemotherapy, these cells will be thawed and given to the subject. . This is called hematopoietic stem cell transplant (HSCT). The final stage of treatment, called maintenance, consists of a drug taken by mouth for 6 months.

Surgery to remove large, or bulky, tumors is a standard part of treatment for high risk neuroblastoma. A few children can have their main tumor removed before chemotherapy, but most require the tumor to shrink first. Surgery has usually been scheduled for after 3 to 5 cycles of therapy, but no one really knows how quickly the tumors are ready to come out. Because chemotherapy has significant side effects that can change the risks of surgery, we will study how early surgeries to remove tumors can happen.

This study is being done to evaluate the outcomes of disease response and survival in children with high risk neuroblastoma treated on this regimen.

DETAILED DESCRIPTION:
Induction Phase Overview The induction phase is approximately 15 weeks long. Chemotherapy is generally given every 3 weeks, each 3 week block is called a "cycle". During these 15 weeks we will treat subjects with chemotherapy 5 times using combinations of 4 different chemotherapy drugs. All IV chemotherapy drugs will be given in the hospital. During this 15 weeks doctors will try to collect special blood cells called hematopoietic stem cells. If the subject's tumor has not been removed completely you will have a surgery to take the rest of the tumor out as soon as possible once it has shrunk with the first two cycles of chemotherapy.

Induction Phase Chemotherapy During the first 2 cycles of chemotherapy all children will receive two drugs: cisplatin and etoposide. Cisplatin is given through an IV for everyone. If participating in the research treatment plan, etoposide by mouth mouth for 14 days. After the first two cycles we will repeat studies to see if the tumor has shrunk. Then all children will receive two other chemotherapy drugs called cyclophosphamide and adriamycin during the 3rd cycle. If the subject responded to the first two cycles, the 4th cycle will be IV cisplatin and oral etoposide again; if the subject did not respond to the first two cycles, the 4th cycle will be IV cisplatin with standard IV etoposide. The 5th cycle will again be adriamycin and cyclophosphamide.

If subjects choose not to participate in the research treatment plan, or are not eligible for the research treatment plan, cycle 1, 2, and 4 will be IV Cisplatin and IV Etoposide.

Here is the induction treatment:

Treatment #1, 2, and 4:

Cisplatin and etoposide: Cisplatin will be given once a day for 5 days through an IV. Etoposide will be given either by mouth once a day for 14 days (research treatment plan) or through an IV for 3 days (standard treatment plan).

Treatment #3 and 5: Cyclophosphamide and adriamycin: Cyclophosphamide and adriamycin are given daily for 2 days, both drugs are given through an IV. Cyclophosphamide may cause irritation of the bladder so another drug called mesna will be given several times after each dose to help prevent this.

After treatment #3 and #5 patients will receive a drug called G-CSF. It stimulates the body to make white blood cells (infection fighting cells) to help prevent infections that can happen because of chemotherapy. G-CSF is an injection that must be given daily.

Surgery: If the primary tumor was not removed before chemotherapy,subjects will undergo a second surgery after receiving chemotherapy. Tumor reevaluation is after cycle #2 and if it is resectable subjects will have surgery at that time. If this is not possible images of the tumor will be taken after cycle #3 and again after cycle #5. Surgery will occur as soon as the tumor is resectable

Stem Cell Harvest Stem cells are special cells that can make all the different types of blood cells. Usually they are found in the bone marrow, but after chemotherapy many more of them are in your blood stream. Between the third and fifth cycles of induction, stem cells will be collected from the blood using a procedure called apheresis. The central line or catheter is connected to a machine that draws some of the subjects blood out of one side of the catheter, filters out the stem cells, and returns the rest of the blood through the other side of the catheter. Each apheresis procedure takes about 4-6 hours. The procedure may need to be done several times to collect enough stem cells.

The consolidation phase takes approximately 15 weeks to complete and consists of radiation to the tumor followed by high doses of chemotherapy and hematopoietic stem cell transplant.

HERE IS THE TREATMENT PLAN:

Local Tumor Radiation:

Local radiation therapy is given daily for about 2 weeks. Radiation beams will be aimed at the sites of the tumor. Each child's treatment will be designed just for them. The doctor who gives radiation will discuss the therapy in detail. Some children require sedation for radiation therapy. Radiation therapy does not usually require admission to the hospital.

High Dose Chemotherapy and Hematopoietic Stem Cell Transplant Carboplatin, etoposide and melphalan: Carboplatin and etoposide are given daily for 4 days followed by melphalan for 3 days. Stem cells will be infused after chemotherapy.

After high dose therapy subjects will receive G-CSF to help stimulate the growth of white blood cells. Other drugs will be used during and after the chemotherapy to prevent or decrease side effects from this treatment. Until the stem cells restore safe levels of blood cells, subjects will need to be hospitalized. This treatment may require hospitalization for 3 to 4 weeks or longer.

Maintenance Phase Starting approximately 3 months following stem cell transplant subjects will receive six monthly treatments with 13-cis-retinoic acid. 13-cis retinoic acid is a drug closely related to vitamin A and has been shown to help stop the multiplication of any remaining neuroblastoma cells in the body. This drug will be taken 2 times a day by mouth for 14 days and then not take it for the following 14 days. This 28-day cycle will be repeated 6 times.

AFTER COMPLETING STUDY TREATMENT The consolidation phase of treatment for high risk neuroblastoma lasts about 4 months. The entire treatment will last about 12-14 months.

ELIGIBILITY:
Inclusion Criteria:

Pts can be enrolled but receive standard etoposide bolus dosing based on clinical conditions at diagnosis (need for emergency intervention because of renal, neurologic, or airway compromise). Pts who meet all other eligibility criteria may also choose to participate in the clinical trial w/o receiving the upfront window protracted dosing of etoposide; these children will receive standard etoposide bolus dosing.

Less than 18 yo at diagnosis

DIAGNOSIS Neuroblastoma or ganglioneuroblastoma verified by histology and/or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites.

Pts with newly diagnosed neuroblastoma and age 365 or more days with the following: * INSS Stage 2a/2b with MYCN amplification , AND unfavorable pathology * INSS Stage 3 with MYCN amplification AND/OR unfavorable pathology

Pts with newly diagnosed neuroblastoma with INSS Stage 4 are eligible with the following: * Age more than 18 months (greater than 547 days) regardless of biologic features * Age 12 to 18 months (365-547 days) with any unfavorable biologic feature (MYCN amplification, unfavorable pathology and/or DNA index equal to 1) or any biologic feature that is indeterminant/unsatisfactory/unknown.

Pts with newly diagnosed neuroblastoma and age less than 365 days with INSS Stage 3, 4, 4S neuroblastoma with MYCN amplification (more than 10).

Pts 365 days or more initially diagnosed with INSS stage 1, 2, 4S who develop distant metastatic disease (meet criteria for INSS stage 4).

Pts may have had no prior systemic therapy except:

* Localized emergency radiation to sites of life threatening or function-threatening disease
* No more than one cycle of chemotherapy according to the intergroup low or intermediate risk neuroblastoma studies prior to determination of MYCN amplification and histology.

TIME FROM DIAGNOSIS Pts must be entered on this study - Within 3 weeks of diagnosis - After recovery from only 1 cycle of chemo on low/intermediate risk NB therapy, - Within 3 weeks of progression with widely metastatic tumor for INSS stage 1, 2, 4S if they received no prior chemotherapy.

HEMATOPOIETIC FUNCTION

* ANC 750/µL or more
* Plt 75,000/µL or more
* or bone marrow involvement with tumor.

LIVER FUNCTION Pts must have adequate liver function defined as

* Direct Bilirubin 1.5 mg/dL or less
* AST and ALT 5 x ULN or less

Pts of childbearing potential must practice an effective method of birth control while on study.

Exclusion Criteria:

Patients who do not meet inclusion criteria.

Patients who are pregnant or lactating are not eligible.

EXCLUSION CRITERIA UPFRONT WINDOW Patients can be enrolled onto Stratum 1 but receive standard etoposide bolus dosing based on clinical conditions at diagnosis. Patients who meet all other eligibility criteria may also choose to participate in the clinical trial without receiving the upfront window protracted dosing of etoposide; these children will receive standard etoposide bolus dosing.

Patients whose tumor requires emergency intervention because of spinal cord compression, CNS compromise, or airway compromise.

Patients requiring dialysis.

If the patient and/or the patient's legally authorized guardian chose to participate in the clinical trial but chose to not participate in the phase II upfront window.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-03; Primary Completion 2009-07 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zage, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase II Window With Protracted Etoposide: 2 cycles of induction therapy for patients who received the Phase II window with Protracted Etoposide
- Phase II Window With Bolus Etoposide: 2 cycles of induction therapy for patients who received the Phase II window with Bolus Etoposide
Period: Overall Study
Arm/Group | Phase II Window With Protracted Etoposide | Phase II Window With Bolus Etoposide
Started | 7 | 6
Completed | 6 (died of complications of surgery after 2 cycles) | 6
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase II Window With Protracted Etoposide | Phase II Window With Bolus Etoposide | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Median (Full Range); unit: month] | 26.9 [17.7 to 130.8] | 25.3 [8.4 to 34.3] | 26.9 [8.4 to 130.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Response Rate Associated With Two Cycles of Cisplatin With Protracted Oral Etoposide When Administered as Up-front Window Therapy to Previously Untreated Children With High Risk Neuroblastoma Tumors.
Description: Partial response or better
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Window With Protracted Etoposide | Phase II Window With Bolus Etoposide
Number analyzed (Participants) | 7 | 6
Participants | 1 | 2
Statistical Analysis 1: Comparison: Phase II Window With Protracted Etoposide vs Phase II Window With Bolus Etoposide; Test type: Superiority or Other; p = 0.367, Fisher Exact

2. Primary Outcome: Rate of Toxicities Associated With Cisplatin With Protracted Oral Etoposide When Administered as Up-front Window Therapy to Previously Untreated Children With High Risk Neuroblastoma.
Description: If a patient experiences any one of the following toxicities, attributed to induction chemotherapy cycles 1, or 2, that patient will be counted as having a dose limiting toxicity. 13.2.1.1 Inability to achieve ANC > 750 by Day 35 from start of chemotherapy cycle 1 or 2 (unless documented tumor involvement of marrow) 13.2.1.2 Inability to achieve platelet count at least 75,000 by Day 35 from start of chemotherapy cycle 1 or 2 (unless documented tumor involvement of marrow) 13.2.1.3 Any Grade 2 or greater toxicity non-hematopoietic/non-mucosal (mucositis/stomatitis) that is not reversible to Grade 1 or baseline by day 21 from start of chemotherapy cycle excluding Hematopoietic toxicity Mucositis/stomatitis Anorexia, nausea, vomiting Febrile neutropenia
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Window With Protracted Etoposide | Phase II Window With Bolus Etoposide
Number analyzed (Participants) | 7 | 6
Participants | 0 | 0

3. Secondary Outcome: Overall Survival in Children With High Risk Neuroblastoma Treated on This Regimen.
Time Frame: 3 years
Population: number of survival
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Window With Protracted Etoposide | Phase II Window With Bolus Etoposide
Number analyzed (Participants) | 7 | 6
Participants | 3 | 2

4. Secondary Outcome: Number of Patients Who Have Surgery After the Second Cycle of Induction Therapy
Description: the measure is the number of patients who have surgery after two cycles of induction
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Window With Protracted Etoposide | Phase II Window With Bolus Etoposide
Number analyzed (Participants) | 7 | 6
Participants | 4 | 2
Statistical Analysis 1: Comparison: Phase II Window With Protracted Etoposide vs Phase II Window With Bolus Etoposide; Test type: Superiority or Other; p = 0.592, Fisher Exact

5. Secondary Outcome: Event Free Survival in Children With High Risk Neuroblastoma Treated on This Regimen.
Description: The first of the two events (relapse or death) was chosen to represent disease free survival
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Window With Protracted Etoposide | Phase II Window With Bolus Etoposide
Number analyzed (Participants) | 7 | 6
Participants | 2 | 1

ADVERSE EVENTS:
Arm/Group | Phase II Window With Protracted Etoposide | Phase II Window With Bolus Etoposide
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II Window With Protracted Etoposide (N=7) | Phase II Window With Bolus Etoposide (N=6)
Allergic reaction to Caspofungin (Immune system disorders) | 1 (1) | 0 (0)
Hearing- monitoring program (Ear and labyrinth disorders) | 1 (1) | 1 (1)
ALC (Blood and lymphatic system disorders) | 2 (9) | 0 (0)
ANC (Blood and lymphatic system disorders) | 7 (44) | 6 (45)
Hemoglobin (Blood and lymphatic system disorders) | 7 (47) | 6 (27)
PLT (Blood and lymphatic system disorders) | 7 (58) | 6 (56)
WBC (Blood and lymphatic system disorders) | 6 (28) | 6 (39)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Hypoxia (Cardiac disorders) | 1 (1) | 0 (0)
INR (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
PTT (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Rash- dermatitis assoc XRT (foot) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ascites, non-malignant (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis/stomatitis (Gastrointestinal disorders) | 2 (2) | 5 (5)
Oral Mucositis/stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage/bleeding abdomen (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Infections and infestations) | 7 (12) | 6 (10)
Infection (Infections and infestations) | 2 (3) | 1 (1)
Infection w/ grade 3 neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Infection w/ grade 4 neutropenia (Infections and infestations) | 1 (2) | 1 (1)
Infection w/Grade2 ANC (Infections and infestations) | 1 (1) | 0 (0)
Infection w/grade 3 ANC (Infections and infestations) | 2 (3) | 2 (2)
Infection w/grade 3/4 ANC (Infections and infestations) | 1 (2) | 1 (1)
Infection w/grade 4 ANC (Infections and infestations) | 3 (3) | 5 (11)
Infection w/normal ANC (Infections and infestations) | 4 (6) | 2 (4)
Infection w/unknown ANC (suspected yeast) (Infections and infestations) | 0 (0) | 1 (1)
Infection with Gr 3/4 neutropenia (candida) (Infections and infestations) | 1 (1) | 0 (0)
Syphillis (Infections and infestations) | 1 (1) | 0 (0)
edema-trunk (Infections and infestations) | 0 (0) | 1 (1)
ALT (Metabolism and nutrition disorders) | 2 (4) | 2 (3)
AST (Metabolism and nutrition disorders) | 2 (4) | 3 (3)
Acidosis (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Bicarbonate (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
GGT (Metabolism and nutrition disorders) | 5 (6) | 5 (7)
Hemoglobin (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 5 (11) | 4 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 4 (6)
Sodium (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Somnolence/depressed lvl consc. (Nervous system disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Infection with normal ANC (parainfluenza) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Vessel Injury/hepatic splenic arteries (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes